CLINICAL TRIAL: NCT00469209
Title: Phase I/II Study of the Combination of Bortezomib With Arsenic Trioxide, Ascorbic Acid and High-Dose Melphalan for Patients With Multiple Myeloma
Brief Title: Velcade, Trisenox, Vitamin C and Melphalan for Myeloma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0893
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2011-04-25 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Myeloma
Keywords: Multiple Myeloma; Melphalan; Trisenox; Arsenic Trioxide; Ascorbic Acid; Vitamin C; Velcade; Bortezomib
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Arsenic Trioxide; Bortezomib; Melphalan; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Bortezomib (Active Comparator): Arm 1: Melphalan 100 mg/m^2 intravenous (IV) days -4,-3 + Arsenic Trioxide 0.25 mg/kg IV for 7 days + Vitamin C IV daily
  Interventions: Drug: Trisenox (Arsenic Trioxide); Drug: Melphalan; Drug: Vitamin C (Ascorbic Acid)
- Bortezomib 1.0 mg/m^2 (Active Comparator): Arm 2: Bortezomib (Level 1) 1.0 mg/m^2 IV push on Days -9, -6, and -3, Melphalan 100 mg/m^2 IV days -4,-3 + Arsenic Trioxide 0.25 mg/kg IV for 7 days + Vitamin C IV daily
  Interventions: Drug: Trisenox (Arsenic Trioxide); Drug: Velcade (Bortezomib); Drug: Melphalan; Drug: Vitamin C (Ascorbic Acid)
- Bortezomib 1.5 mg/m^2 (Active Comparator): Arm 3: Bortezomib (Level 2) 1.5 mg/m^2 IV push on Days -9, -6, and -3, Melphalan + Arsenic Trioxide 0.25 mg/kg IV for 7 days + Vitamin C IV daily
  Interventions: Drug: Trisenox (Arsenic Trioxide); Drug: Velcade (Bortezomib); Drug: Melphalan; Drug: Vitamin C (Ascorbic Acid)

INTERVENTIONS:
Drug: Trisenox (Arsenic Trioxide) — 0.25 mg/kg by vein over 2 hours, once a day for 7 days (Days -9 to -3).
  Other Names: ATO
Drug: Velcade (Bortezomib) — Arm 1 (Level 1):
  1.0 mg/m^2 intravenous (IV) push on Days -9, -6, and -3. An IV push takes a short period of time (less than 1 minute).
  Arm 2 (Level 2):
  1.5 mg/m^2 intravenous (IV) push on Days -9, -6, and -3. An IV push takes a short period of time (less than 1 minute).
  Other Names: PDP-341; MLN341; PS-341
  Arms: Bortezomib 1.0 mg/m^2; Bortezomib 1.5 mg/m^2
Drug: Melphalan — 100 mg/m2 by vein days -4,-3, over 30 minutes
  Other Names: Alkeran
Drug: Vitamin C (Ascorbic Acid) — 1000 mg once a day through the vein for 7 days.

SUMMARY:
Primary Objectives:

1. To evaluate the toxicity and safety of a combination of bortezomib with arsenic trioxide, ascorbic acid and high-dose melphalan in patients with multiple myeloma
2. To evaluate the efficacy of a combination of bortezomib with arsenic trioxide, ascorbic acid and high-dose melphalan in patients with multiple myeloma
3. To determine the effects of bortezomib on melphalan pharmacokinetics

DETAILED DESCRIPTION:
Melphalan is designed to damage the DNA of cells, which may cause cancer cells to die. High-dose melphalan is considered the standard of care for multiple myeloma. Bortezomib is designed to block a protein that plays a role in cell function and growth, which may cause cancer cells to die. Arsenic trioxide may cause cancer cells to die, and researchers want to find out if arsenic trioxide helps melphalan in killing cancer cells. Vitamin C makes arsenic trioxide more available inside the cancer cells, and researchers want to learn if Vitamin C makes arsenic trioxide more effective.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate). Your complete medical history will be recorded. You will have a dental exam to check for any infected teeth or gums that may flare up after chemotherapy.

You will have a bone marrow aspirate and biopsy. To collect a bone marrow aspirate/biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle. Cytogenetic tests will be performed on the aspirate sample to look for any genetic abnormalities in your DNA. You will have x-rays of your bones taken. The study doctor will look at the x-rays to see if there are any myeloma-related bone changes. You will also have a chest x-ray.

You will have blood (about 2 tablespoons) and urine collected for routine tests. You will have a pulmonary function test, to check if your lungs are strong enough for high-dose chemotherapy. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). You will also have a MUGA scan to evaluate the function of your heart. Women who are able to have children must have a negative blood pregnancy test. The blood will be drawn as part of the 2 tablespoons drawn at screening.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of dice) to one of 3 treatment groups. There is an equal chance of being assigned to any of the 3 groups. All 3 groups will receive melphalan, arsenic trioxide, and Vitamin C. The second and third groups will also receive bortezomib, but at different dose levels. The first 3 participants assigned to receive bortezomib on this study will receive the lower of 2 bortezomib dose levels.

You will receive arsenic trioxide through a needle in a vein over 2 hours, once a day for 7 days (Days -9 to -3). At the same time, you will receive Vitamin C once a day through the vein for 7 days. After you receive the arsenic trioxide on Days -4 and -3, you will receive melphalan through the vein over 30 minutes.

If you are in Group 2 or 3, you will receive bortezomib by an intravenous (IV) push on Days -9, -6, and -3. An IV push takes a short period of time (less than 1 minute).

You will receive standard inpatient and outpatient stem cell transplant care and testing. You will have to sign a separate consent form that describes the transplant procedure and its risks. Your stem cells will be reinfused 2 days after the last dose of melphalan. To check for any side effects, you will have an ECG performed 14 days after the transplant.

If intolerable side effects from the chemotherapy occur or there is sign of disease after the transplant, you will be taken off study. If you have already received melphalan and side effects occur, then the transplant will happen. However, if intolerable side effects develop before melphalan, then you may be taken off study without having the transplant. If you are taken off study early, you still may need to return for routine post-transplant follow-up visits, if your transplant physician decides it is necessary.

If there is no sign of disease after the transplant, you will have routine follow-up visits. Blood (about 2 tablespoons) will be drawn for routine tests at least once a week during the first month after the transplant, and then once every month for the next 3 months after that. At about 3, 6, and 12 months after the transplant, you will have bone marrow biopsies and aspirates performed to check the status of the disease. You will have blood (about 2 tablespoons) and urine collected for routine tests. At 12 months after the transplant, you will have x-rays of your bones taken.

One (1) year after the transplant, your participation in this study will be over.

This is an investigational study. Bortezomib, arsenic trioxide, and melphalan are commercially available and FDA-approved for use in patients with myeloma. However, their use in combination with Vitamin C (also commercially available) is investigational. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. a) Primary Refractory Disease (defined as failure to achieve even a partial response to induction therapy) b) Consolidation of a partial remission (defined as a decrease but continued presence of monoclonal protein on serum and urine immunofixation electrophoresis, and/or the presence of plasmacytosis on bone marrow aspirate and biopsy) c) Relapsing after prior therapy (disease relapsing after achieving a partial or complete response to prior conventional or high-dose therapy).
2. Age up to 75 years.
3. Zubrod performance status of <2.
4. Left ventricular ejection fraction >40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
5. Forced expiratory volume (FEV1), forced volume vital capacity (FVC) and Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) >40%. No symptomatic pulmonary disease.
6. Serum bilirubin <2 times upper limit of normal, alanine aminotransferase/SGPT <4 times upper limit of normal. No evidence of chronic active hepatitis or cirrhosis. No effusion or ascites >1L prior to drainage.
7. HIV-negative.
8. Negative Beta human chorionic gonadotrophin (hCG) test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization
9. Patient or guardian able to sign informed consent
10. Corrected QT interval less than 470 msec.

Exclusion Criteria:

1. Corrected QT interval greater than 470 msec.
2. Patients in complete remission (defined as the absence of monoclonal protein on serum and urine immunofixation electrophoresis, and the absence of plasmacytosis in bone marrow aspirate and biopsy).
3. Patients with non-secretory myeloma.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H. Qazilbash, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period June 2006 to December 2008. All participants recruited at UT MD Anderson Cancer Center.
Groups:
- No Bortezomib: Melphalan 100 mg/m^2 intravenous (IV) days -4,-3 + Arsenic Trioxide 0.25 mg/kg IV for 7 days + Vitamin C IV daily
- Bortezomib 1.0 mg/m^2: Bortezomib (Level 1) 1.0 mg/m^2 IV push on Days -9, -6, and -3, Melphalan 100 mg/m^2 IV days -4,-3 + Arsenic Trioxide 0.25 mg/kg IV for 7 days + Vitamin C IV daily
- Bortezomib 1.5 mg/m^2: Bortezomib (Level 2) 1.5 mg/m^2 IV push on Days -9, -6, and -3, Melphalan + Arsenic Trioxide 0.25 mg/kg IV for 7 days + Vitamin C IV daily
Period: Overall Study
Arm/Group | No Bortezomib | Bortezomib 1.0 mg/m^2 | Bortezomib 1.5 mg/m^2
Started | 20 | 20 | 20
Completed | 19 | 20 | 19
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Bortezomib | Bortezomib 1.0 mg/m^2 | Bortezomib 1.5 mg/m^2 | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 70] | 59 [45 to 67] | 64 [49 to 75] | 60 [45 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 6 | 27
  Male | 8 | 11 | 14 | 33
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reaching Complete Response (CR)
Description: Number of participants with CR at Day 180 who had maintained CR for at minimum of 4 weeks, and who had: No monoclonal protein in urine/serum when analyzed by immunofixation electrophoresis; bone marrow normal by morphological examination with <5% plasma cells, <1% aneuploid light chain restricted population by flow cytometry for DNA/cIg; and, while healing of bony lesion is not required, no new lytic lesion should appear. Further compression fracture of spine not considered progressive disease.
Time Frame: Baseline through Day 180, with assessments at Day 90 and Day 180
Population: Analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | No Bortezomib | Bortezomib 1.0 mg/m^2 | Bortezomib 1.5 mg/m^2
Number analyzed (Participants) | 20 | 20 | 20
participants | 4 | 1 | 4

2. Secondary Outcome: Time to Toxicity
Description: The time to patient toxicity of drug combination bortezomib with arsenic trioxide, ascorbic acid and high-dose melphalan defined in days from baseline measure to occurence of adverse events grade 4 (life threatening or disabling) according to National Cancer Institute Common Toxicity Criteria (CTC), version 3.
Time Frame: Baseline to event occurence (assessed weekly first 30 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study period 2 years.
Arm/Group | No Bortezomib | Bortezomib 1.0 mg/m^2 | Bortezomib 1.5 mg/m^2
Serious Adverse Events (participants affected / at risk) | 3/20 | 2/20 | 2/20
Other Adverse Events (participants affected / at risk) | 4/20 | 5/20 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Bortezomib (N=20) | Bortezomib 1.0 mg/m^2 (N=20) | Bortezomib 1.5 mg/m^2 (N=20)
pneumonitis/death (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ventriculat tachycardia/hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Bortezomib (N=20) | Bortezomib 1.0 mg/m^2 (N=20) | Bortezomib 1.5 mg/m^2 (N=20)
mucositis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
low back pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
elevated transaminases (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No